CLINICAL TRIAL: NCT03657966
Title: An Open-label, Single-group, Multi-center, Phase II Clinical Trial Evaluating the Effect of Maintenance DCVAC/OvCa After Standard-of-care Therapy in Women With First Relapse of Platinum-sensitive Epithelial Ovarian Cancer
Brief Title: DCVAC/OvCa After Standard-of-care Chemotherapy in Women With Relapse of Platinum-sensitive Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOV06; 2017-002196-26 (EudraCT Number)
Record Dates: First submitted 2018-08-24; First posted 2018-09-05 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Ovarian Cancer Recurrent
Keywords: Immunotherapy; Platinum-sensitive; Biologic; Vaccine; Ovarian cancer; Fallopian Tube cancer; Primary peritoneal cancer; dendritic cells; chemotherapy; leukapheresis; FIGO III; FIGO IV
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin; Gemcitabine; Paclitaxel

STUDY DESIGN:
Intervention Model Description: open-label DCVAC/OvCa after treatment with carboplatin in combination with either gemcitabine or paclitaxel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard of care chemotherapy + DCVAC/Ov (Experimental): Standard-of-care carboplatin/gemcitabine or carboplatin/paclitaxel followed by DCVAC/OvCa
  Interventions: Biological: DCVAC/OvCa; Drug: Standard of Care Chemotherapy

INTERVENTIONS:
Biological: DCVAC/OvCa — activated dendritic cells (DCVAC/OvCa) for immune maintenance after chemotherapy
Drug: Standard of Care Chemotherapy — either carboplatin and gemcitabine or carboplatin and paclitaxel followed by DCVAC/OvCa
  Other Names: carboplatin with gemcitabine; carboplatin with paclitaxel

SUMMARY:
The purpose of this trial is to investigate if maintenance DCVAC/OvCa after second-line chemotherapy of carboplatin/gemcitabine or carboplatin/paclitaxel improves efficacy outcomes in women with FIGO stage III and IV epithelial ovarian carcinoma who experienced relapse more than 6 months after complete remission of first line platinum-based chemotherapy (platinum sensitive ovarian cancer)

DETAILED DESCRIPTION:
All patients who fulfill all eligibility criteria will undergo a leukapheresis procedure. All eligible/enrolled patients will receive standard-of-care therapy with carboplatin/gemcitabine or carboplatin/paclitaxel starting 2 to 7 days after leukapheresis.

After 6 cycles of chemotherapy, patients will start maintenance treatment with DCVAC/OvCa.

Treatment will continue irrespective of tumor progression until completion, refusal, intolerance of treatment or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed FIGO stage III or IV epithelial ovarian, primary peritoneal or fallopian tube carcinoma (serous,endometrioid, or mucinous) who had complete remission after first-line platinum-based chemotherapy
* Radiologically confirmed relapse after >6 months of remission ( platinum-sensitive cancer)
* Laboratory parameters per protocol

Exclusion Criteria:

* FIGO I, II epithelial ovarian cancer
* FIGO III, IV clear cells epithelial ovarian cancer
* Non-epithelial ovarian cancer
* Borderline tumors ( tumors of low malignant potential)
* Prior or current systemic anti-cancer therapy for ovarian cancer (chemotherapy, monoclonal antibody therapy, tyrosine kinase inhibitory therapy, vascular endothelial growth factor or hormonal therapy) except first-line Pt based chemotherapy ( with or without bevacizumab)
* fertile women of child-bearing potential not willing to use a highly effective method of contraception or a combination of methods
* Pregnant of lactating women
* Pre-defined co-morbidities
* Known hypersensitivity to any constituent of DCVAC/OVCa or the selected chemotherapy compounds

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 33 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival by modifications to the RECIST 1.1 | Assessed from enrollment up to 104 weeks
  PFS as defined as the time from the first dose of Standard-of-Care (SoC) therapy administerd until tumor progression or death from any cause

SECONDARY OUTCOMES:
Overall survival | Assessed from enrolment through study completion approximately 5 years
  Defined as the time from first dose of SoC therapy administered until death due to any cause assessed until study completion
Biological progression-free interval | CA-125 assessed every 6 weeks up to 104 weeks
  Defined by increasing CA-125 levels per Gynecologic Cancer Intergroup (GCIG) criteria
Objective Response rate | Response is assessed every 8 weeks up to 104 weeks
  CR and PR measured by the modifed RECIST 1.1 criteria
Immunologic Response | Blood samples collected 5 times throughout the study from enrolment up to 104 weeks
  Detection of entire anti-tumor immune response int he serum
Incidence of Treatment-emergent adverse events [safety and tolerability] | Screening through 30 days after completion of treatment
  Safety profile as determined by the nature, incidence, duration, severity and outcome of adverse events (AEs) including serious AEs (SAEs) as assessed by CTCAE v. 4.0
CA-125 response | CA-125 assessed every 6 weeks up to 104 weeks
  Defined by GCIG criteria
Time to either tumor or biologic Response | From first dose of chemotherapy until either objective or serologic progression for up to 104 weeks.
  Response according to RECIST or CA-125 measurements as increased to >2 times ULN

CONTACTS AND LOCATIONS:
Overall Officials: Harald Fricke, MD, PhD, Study Director — SOTIO a.s.
Locations (8):
- Czechia (8):
  - University Hospital Brno, Brno
  - Masaryk Memorial Cancer Institute, Brno
  - Hospital Novy Jicin, Nový Jičín
  - University Hospital in Ostrava, Ostrava
  - University Hospital Plzen, Pilsen
  - University Hospital Kralovsko Vinohrady, Prague
  - General University Hospital in Prague, Prague
  - Hospital Bulovka, Prague

IPD SHARING:
Plan to Share IPD: Undecided